CLINICAL TRIAL: NCT04567173
Title: A Randomized, Open-Label, Single Center Clinical Trial to Assess the Efficacy and Safety of Convalescent Plasma to Hospitalized Adult COVID-19 Patients as Adjunctive Therapy to Reduce the Need for ICU Admission: Co-CLARITY Trial
Brief Title: Convalescent Plasma as Adjunctive Therapy for Hospitalized Patients With COVID-19
Acronym: Co-CLARITY
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Limited enrolment (unable to achieve target sample size)
Sponsor: University of the Philippines (Other)
Responsible Party: Principal Investigator, Deonne Thaddeus Gauiran, Principal Investigator, University of the Philippines
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PHRR200824-002868
Record Dates: First submitted 2020-09-24; First posted 2020-09-28 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Covid19
Keywords: COVID-19; Convalescent plasma
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: This is a phase 3, randomized, non-placebo controlled, open-label, non-blinded, single-center clinical trial which will assess the efficacy and safety of anti-SARS-CoV-2 convalescent plasma given from the 3rd to 14th day of illness after the onset of symptoms in preventing ICU admission among COVID-19 patients compared to standard of care. Consequently enrolled patients will be randomized using the REDCap randomization module
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anti-SARS-CoV-2 convalescent plasma (Experimental): About 500 mL of type-specific anti-SARS-CoV-2 convalescent plasma collected by whole blood donation or standard pheresis from a volunteer who recovered from COVID-19 transfused intravenously as 2 aliquots of 250 mL
  Interventions: Drug: Anti-SARS-CoV-2 convalescent plasma
- Standard of care (No Intervention): Patients in the control group are those will only receive local standard of care as deemed appropriate by the primary attending physicians and guided by institutional pathways

INTERVENTIONS:
Drug: Anti-SARS-CoV-2 convalescent plasma — convalescent plasma derived from whole blood donors or standard pheresis from a volunteer who recovered from COVID-19
  Arms: Anti-SARS-CoV-2 convalescent plasma

SUMMARY:
This protocol provides access to investigational convalescent plasma for hospitalized patients with COVID-19. Following provision of informed consent, patients will be administered around 500 mL of convalescent plasma obtained from an individual who has recovered from a documented SARS-CoV-2 infection. The study aims to evaluate the efficacy and safety of anti-SARS-CoV-2 convalescent plasma as adjunctive therapy in preventing disease progression (prevention of ICU admission) among hospitalized patients with COVID-19. Safety outcomes include serious adverse events judged to be related to convalescent plasma. Other information which will be collected includes patient demographics and clinical data which includes quick SOFA scores, ventilator-free days, ICU-free days, dialysis-free days and 28-day mortality.

DETAILED DESCRIPTION:
This is a phase 3, randomized, non-placebo controlled, open-label, single-center clinical trial which will assess the efficacy and safety of anti-SARS-CoV-2 convalescent plasma given from the 3rd to 14th day of illness after the onset of symptoms in preventing ICU admission among hospitalized COVID-19 patients compared to standard of care. Consecutive patients with COVID-19 admitted to the UP Philippine General Hospital will be offered participation into the study. Patients in the intervention group will receive one dose of type-specific anti-SARS-CoV-2 convalescent plasma (500 mL collected by whole blood donation or standard pheresis at the UP-PGH blood bank from a volunteer who recovered from COVID-19). The primary safety endpoints include serious adverse events judged to be related to convalescent plasma. The study also aims to compare anti-SARS-CoV-2 antibody titers and rates, levels, and duration of SARS-CoV-2 RNA in nasopharyngeal swabs using RT-PCR between the intervention and control groups.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be 19 years of age or older
* Hospitalized with COVID-19 and confirmed via SARS-CoV-2 RT-PCR testing
* Patient is willing and able to provide written consent and comply with all protocol requirements
* Patient agrees to storage of specimens for future testing

Exclusion Criteria:

* Female subjects with positive pregnancy test, are breastfeeding or planning to become pregnant/breastfeed during the study period
* Symptomatic illness exceeding 14 days from onset of illness at time of enrollment
* ICU admission on initial presentation at the hospital (includes patients with clinical indications for ICU admission as follows:

  1. Respiratory distress with requirement of O2 >6 lpm to maintain O2 sat >92%
  2. Rapid escalation of O2 requirement/significant work of breathing
  3. Hemodynamic instability: SBP <90, MAP <65
* Receipt of any blood products including pooled immunoglobulin or intravenous immunoglobulin (IVIg) in the past 30 days prior to enrolment
* Known IgA deficiency
* Presence of any contraindication to transfusion (or history of prior severe reactions to transfusion of blood products)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2020-09-21 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Incidence of serious adverse events | 28 days from enrollment
  Cumulative incidence of serious adverse events (transfusion-related acute lung injury, transfusion associated circulatory overload, transfusion related infection and anaphylaxis/severe allergic reactions) during the study period

SECONDARY OUTCOMES:
Quick SOFA (qSOFA) score | 28 days from enrollment
  Quick Sequential Organ Failure Assessment (qSOFA) scores of study participants within 28 days from enrollment. The qSOFA score is a rapid bedside clinical score used to identify patients with suspected infection that are at a greater risk for a poor outcome. Minimum score is 0 and maximum score is 3. A higher score is associated with higher risk for in-hospital mortality.
Cardiopulmonary arrest | 28 days from enrollment
  Total number of patients experiencing cardiopulmonary arrest
ICU mortality | 28 days from enrollment
  Total number of deaths among patients admitted to the ICU
ICU length of stay | 28 days from enrollment
  Total number of days patients were admitted to the ICU
Hospital mortality | 28 days from enrollment
  Total number of deaths among study participants
Hospital length of stay | 28 days from enrollment
  Total number of days patients were admitted to the hospital
Dialysis-free days | 28 days from enrollment
  Days without dialysis within 28 days from enrollment
Vasopressor-free days | 28 days from enrollment
  Days without vasopressors within 28 days from enrollment
ICU-free days | 28 days from enrollment
  Days without need for ICU admission within 28 days from enrollment
28-day mortality | 28 days from enrollment
  Total number of patient deaths within 28 days from enrollment
Anti-SARS-CoV-2 antibody titers | days 0, 1, 7 and 14 of enrollment
  Anti-SARS-CoV-2 IgG antibody titers
SARS-CoV-2 RNA by RT-PCR | days 0, 1, 7 and 14 of enrollment
  Levels of SARS-CoV-2 RNA in nasopharyngeal swabs (or other specimen types as available) using RT-PCR

CONTACTS AND LOCATIONS:
Overall Officials: Deonne Thaddeus V Gauiran, MD, Principal Investigator — UP Philippine General Hospital
Locations (1):
- UP Philippine General Hospital, Manila, Philippines